CLINICAL TRIAL: NCT02852083
Title: A Prospective Phase II, Randomized Multi-center Trial of a Combined Modularized Treatment With Metronomic Low-dose Treosulfan, Pioglitazone and Clarithromycin Versus Nivolumab in Patients With Squamous Cell Lung Cancer and Non- Squamous Cell Lung Cancer, Respectively After Platin Failure
Brief Title: A Trial With Metronomic Low-dose Treosulfan, Pioglitazone and Clarithromycin Versus Standard Treatment in NSCLC
Acronym: ModuLung
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Regensburg (Other)
Collaborators: The Anticancer Fund (Unknown)
Responsible Party: Principal Investigator, Albrecht Reichle, Prof. Dr., University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ModuLung
Record Dates: First submitted 2016-07-12; First posted 2016-08-02 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Squamous Cell Lung Cancer; Non-Squamous Cell Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pioglitazone; Nivolumab; treosulfan; Clarithromycin

ARMS (2):
- A: Biomodulatory treatment (Experimental): treosulfan 250 mg p.o. twice daily, pioglitazone 45 mg p.o. once daily, clarithromycin 250 mg p.o. twice daily until progression or no clinical benefit observed, whichever comes first.
  Interventions: Drug: Pioglitazone; Drug: Treosulfan; Drug: Clarithromycin
- B: Standard Treatment (Active Comparator): Nivolumab, 3 mg per kilogram of body weight every 2 weeks until disease progression according to RECIST 1.1 or unacceptable toxicity
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 25 mg once daily, p.o.
  Other Names: Actos
  Arms: A: Biomodulatory treatment
Drug: nivolumab — 3 mg per kilogram of body weight every 2 weeks, p.o. (standard treatment)
  Other Names: Opdivo
  Arms: B: Standard Treatment
Drug: Treosulfan — Treosulfan 250 mg twice daily, p.o.
  Arms: A: Biomodulatory treatment
Drug: Clarithromycin — Clarithromycin 250 mg twice daily p.o.
  Arms: A: Biomodulatory treatment

SUMMARY:
This is a Phase II, multicentre, open-label, randomized, and controlled study, evaluating the efficacy and safety of combined modularized treatment of treosulfan, pioglitazone and clarithromycin in patients with with squamous and non- squamous cell lung cancer, respectively after platin failure.

DETAILED DESCRIPTION:
Patients will be randomized 1:1, and will be stratified according to histology (squamous cell carcinoma vs adenocarcinoma).

86 patients with platin refractory Non-Small Cell Lung Cancer (NSCLC) will be treated either with metronomic low-dose treosulfan, pioglitazone and clarithromycin (experimental arm) or with nivolumab (squamous cell lung cancer and nonsquamous cell lung cancer).

Patients will undergo tumor assessments at baseline and every 6 weeks (approximately every two cycles) thereafter, until progression. Patients without progression after 36 weeks will undergo tumor assessments every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Ability to comply with protocol
* Age ≥ 18 years
* Measurable disease, as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Histologically or cytologically confirmed locally advanced or metastatic (i.e., Stage IIIB not eligible for definitive chemoradiotherapy, Stage IV, or recurrent) NSCLC (per the Union Internationale Contre le Cancer/American Joint Committee on Cancer [UICC/AJCC] staging system);
* Disease progression during or following treatment with a prior platinum containing regimen for locally advanced, unresectable/inoperable or metastatic NSCLC or disease recurrence within 6 months of treatment with a platinum based adjuvant/neoadjuvant regimen
* No more than 2 cytotoxic chemotherapy regimens
* Patients that have progressed during or after treatment with EGFR Tyrosine Kinase Inhibitor (TKI) in first line, or are intolerant to treatment with erlotinib, gefitinib, or another EGFR TKI may be included.
* Patients that have progressed during or after , or intolerant to treatment with crizotinib or another ALK inhibitor
* The last dose of prior systemic anti-cancer therapy must have been administered ≥ 21 days prior to randomization (≥ 14 days for vinorelbine or other vinca alkaloids or gemcitabine.)
* The last dose of treatment with any investigational agent must have ended ≥ 28 days prior to randomization.
* Prior radiation therapy is allowed provided recovery from any toxic effects thereof and ≥ 7 days between the last fraction and randomization.
* Adequate hematologic and end organ function, defined by the following (max 14 days prior study treatment): Absolute Neutrophil Count (ANC) ≥ 1500 cells/μL (without granulocyte colonystimulating factor support within 2 weeks of sampling), White Blood Cell (WBC) counts > 2,500/μL and < 15,000/μL, lymphocyte count ≥ 500/μL, Platelet count ≥ 100,000/μL (without transfusion within 2 weeks of sampling), Hemoglobin ≥ 9.0 g/dL. Transfusion or erythropoietic treatment is allowed.
* Liver function tests meeting one of the following criteria: Aspartate Transaminase (AST) or Alanine Transaminase (ALT) ≤ 2.5 × ULN, with normal alkaline phosphatase or AST and ALT ≤ 1.5 × ULN in conjunction with alkaline phosphatase > 2.5 × ULN; Serum bilirubin ≤ 1.0 × ULN. Patients with known Gilbert's disease must have serum bilirubin level ≤ 3 × ULN.
* Prothrombin Time - International Normalized Ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, without anticoagulants. Patients receiving therapeutic anticoagulation must be on a stable dose for at least 1 week prior to randomization.
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for 6 months after the last dose of the combined modularized treatment.
* Patients must have recovered from all acute toxicities from previous therapy, excluding alopecia.

Exclusion Criteria:

Cancer-Specific Exclusion Criteria

* Known active or untreated central nervous system (CNS) metastases.Patients with a history of treated asymptomatic CNS metastases are eligible, if they meet all of the following criteria: No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus. Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
* History of intracranial hemorrhage
* Ongoing requirement for dexamethasone for CNS disease
* Stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1,Day 1
* Screening CNS imaging ≥ 4 weeks since completion of radiotherapy and ≥ 2 weeks since discontinuation of corticosteroids
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression that has not been clinically stable for ≥ 2 weeks prior to randomization
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled tumor-related pain: patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy should be treated prior to enrolment. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain should be considered for loco-regional therapy prior to enrolment.
* Hypercalcemia (Ca > 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continuous bisphosphonate therapy or denosumab. Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and without a history of clinically significant hypercalcemia are eligible.
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with curative outcome

General Exclusion Criteria

* History of idiopathic pulmonary fibrosis (including pneumonitis), history of drug-induced pneumonitis
* Serum albumin < 2.5 g/dL
* Patients with active hepatitis B or hepatitis C. Patients with past Hepatitis B Virus (HBV) infection or resolved HBV are eligible. Patients positive for Hepatitis C Virus (HCV) antibody are eligible only if Polymerase Chain Reaction (PCR) is negative for HCV Ribonucleic Acid (RNA).
* Significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease
* Significant cardiovascular disease, such as myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina.
* Known left ventricular ejection fraction (LVEF) < 40%. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen.
* Tuberculosis
* Severe infections within 4 weeks prior to randomization
* oral or intravenous antibiotics within 2 weeks prior to randomization
* Major surgical procedure within 4 weeks prior to randomization or expected need for a major surgical procedure during the course of the study other than for diagnosis
* Prior treatment with nivolumab
* Grade ≥ 2 peripheral neuropathy as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC AE) v4.0 criteria
* Patients undergoing dialysis or creatinine clearance <30 mL per minute,defined according to Modification of Diet in Renal Disease Study Criteria (MDRD)
* Patients with uncontrolled hypertension (Respiratory rate continuously > 140/90 mm Hg)
* Simultaneous treatment with another investigational agent or simultaneous anticancer treatment outside this trial

Exclusion Criteria Related to Study Drugs

* Heart failure > New York Heart Association (NYHA) 1, QT prolongation, ventricular arrhythmias, torsade de pointes
* Creatinine > 1.5 mg/dL
* chronic hypopotassemia
* HIV infection requiring virostatic therapy
* past or current bladder cancer , patients with risk factors for bladder cancer (such as exposure to aromatic amines or heavy tobacco smokers), or macrohematuria of unknown origin
* Known gastrointestinal disorder, including malabsorption or active gastric ulcer, that might interfere with oral intake and absorption of study medication
* Autoimmune disease, symptomatic interstitial lung disease, systemic immunosuppression, prior therapy with T-cell costimulation or checkpoint targeted agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 6 months after study completion

SECONDARY OUTCOMES:
Overall Survival | up to 6 months after study completion
Duration of Response | up to 6 months after study completion
Number of participants experiencing adverse events related to the study drugs | up to 6 months after study completion
  Safety and Tolerability assessments will include the incidence, nature, and severity of adverse events and laboratory abnormalities graded per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.0). Laboratory safety assessments will include, but are not limited to, the regular monitoring of hematology and blood chemistry
Number of participants experiencing a change in cellular secretome analytics in serum | at screening, at the beginning of each new treatment cycle (each cycle consists of 28 days) and at the end of treatment visit, which will take place within 3 weeks of the last intake of study drug
  To measure the effect on inflammation, angiogenesis and immune response (proteomics, lipidomics) on serum samples
proportion of patients who report a considerable degree of impairment in a respective dimension, i.e. a score value <50 | up to 6 months after study completion
  evaluate and compare patient reported outcomes (PROs) of lung cancer symptoms and patient functioning between treatment arms
proportion of patients who report a considerable degree of impairment in a respective dimension, i.e. a score value <50 | up to 6 months after study completion
  evaluate and compare health-related quality of life (HRQoL) between treatment arms
Comparison of participants tumour response according to (Response Evaluation Criteria in Solid Tumors) RECIST criteria version 1.1 and Peroxisome proliferator-activated receptor gamma (PPAR-γ) expression | Baseline
  tissue microarray for analysis of PPAR-γ expression for each tumour sample will be performed.
description of change in predictive and prognostic exploratory biomarkers for each participant | at screening,at the beginning of each treatment cycle (each treatment cycle consists of 28 days), and at the end of treatment visit, which will take place within 3 weeks of the last intake of study drug
  For patients participating in University Clinic Regensburg only: Secretome analytics (proteomics, lipidomics) will be performed to monitor functions of tumor-associated cellular compartments on serum samples. Serum samples are taken at the beginning of each new treatment cycle. epidermal growth factor receptor (EGFR), K-ras, Anaplastic lymphoma kinase (ALK), and Programmed cell death protein 1 (PD-1) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (9):
  - Onkologische Gemeinschaftspraxis Dres. Wilke/ Wagner/Petzoldt, Fürth, Bavaria
  - Klinikum Kempten Oberallgäu, Immenstadt im Allgäu, Bavaria
  - MVZ am Klinikum GmbH, Passau, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Kliniken Nordoberpfalz AG, Klinikum, Weiden, Bavaria
  - MVZ Weiden GmbH, Weiden, Bavaria
  - St. Antonius-Hospital, Eschweiler, North Rhine-Westphalia
  - Klinik für Innere Medizin, Homburg/Saar, Saarland
  - Krankenhaus Martha-Maria, Halle, Saxony-Anhalt